CLINICAL TRIAL: NCT00624455
Title: Does a Single Preoperative Dose of Gabapentin Reduce Postoperative Tonsillectomy Pain and Subsequent Morphine Requirement in Children?
Brief Title: How Does Gabapentin Affects Post-operative Tonsillectomy Pain?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Robert Purdy, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H07-00265
Record Dates: First submitted 2008-02-18; First posted 2008-02-27 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Post-operative Pain
Keywords: Gabapentin; tonsillectomy; post-operative pain; morphine requirements; randomized double blind; adenotonsillectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): One dose of oral premedication of Gabapentin 10 mg kg-1 given at least 30 but not more than 90 minutes before surgery. Max dose is 600mg.
  Interventions: Drug: Gabapentin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — One dose of oral premedication of Gabapentin 10 mg kg-1 given at least 30 but not more than 90 minutes before surgery. Max dose is 600mg.
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Gabapentin is a medicine that has been used in adults (but not yet in children) to treat pain after surgery. In children it has been used for many years to treat other conditions and has been shown to be very safe.

Removal of tonsils is a common operation with each child experiencing a similar pattern of pain; this makes it good for looking at the effect of pain relieving medicines. In our study each child will get the same operation and medicines, as they would have normally. Before the operation and in a random way, half will get gabapentin and half will get the same syrup but with no gabapentin. Afterwards we will record how much pain the children have and how much of our standard medicine is needed to make them comfortable. We expect both of these results to be lower in the half who received gabapentin. We will also record the amount and type of unwanted effects, both from the gabapentin and from any other pain relief medicines.

DETAILED DESCRIPTION:
Tonsillectomy is one of the most commonly performed children's surgeries and produces a consistent pattern and intensity of pain in the recovery period. These qualities make this surgery ideal for the investigation of pain relieving medications. Adequate analgesia for tonsillectomy in the perioperative period presents a challenge to the anesthetist because opiates, which provide the most effective analgesia, are associated with a high incidence of nausea and vomiting, respiratory depression, and sedation. These effects make recovery from tonsillectomy particularly hazardous in children with Obstructive Sleep Apnea Syndrome (OSAS) (the primary indication for tonsillectomy or adenotonsillectomy) thus alternatives to opiates have been sought. Gabapentin is a drug with an extensive safety record in the treatment of children's seizures, and chronic pain syndromes. Recently studies have demonstrated new modes of action for this medication, both directly on pain and in increasing the efficacy of conventional opiate (morphine) pain relieving medications. As such it may have role in the relief of acute pain. We hypothesize that given preoperatively as a single dose; gabapentin will reduce postoperative pain and opiate requirement in children undergoing tonsillectomy. Randomization will follow a computer generated random pattern with 14 patients in each group (placebo or gabapentin). Pain and sedation will be recorded as will the incidence of vomiting, dizziness and pruritis. Pain will be assessed using the Coloured Analogue Scale and sedation with the University of Michigan Sedation Scale. The time to first oral intake of fluids will also be recorded. All recordings will be made at 5-minute intervals from time of extubation (time = 0) and will be made by an independent blinded recovery nurse. Subjects will stay in the PACU for a minimum of one hour from time zero, and will only be discharged to the Surgical Daycare Unit at a point after this when two successive pain measurements demonstrate a score of 3 or less. In the Surgical Daycare Unit pain assessment will continue at intervals of 30 minutes to a total time of 4 hours from time zero and will be recorded by a member of the research team blinded to nature of premedication. A telephone interview will be scheduled with the subject's parents at 24 hours from time zero.

ELIGIBILITY:
Inclusion Criteria:

* Tonsillectomy
* Adenotonsillectomy
* ASA status 1 to 3
* Weight < 60 kg
* BMI < 30

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Total postoperative morphine consumption at four hours (from the time of extubation) | 4 hours

SECONDARY OUTCOMES:
Pain scores, presence of nausea/ vomiting, dizziness, sedation, satisfaction | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert Purdy, MD, Principal Investigator — University of British Columbia; Mark Ansermino, MD, Study Director — University of British Columbia; Andrew Morrison, MD, Study Director — University of British Columbia; Helen Hume-Smith, MD, Study Director — University of British Columbia; Simon Whyte, MD, Study Director — University of British Columbia; Carolyne Montgomery, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada